CLINICAL TRIAL: NCT06100783
Title: Depot-medroxy Progesterone Acetate Injectable Contraceptives in Lactating Women 1st Week Versus 6 Week Postpartum Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Boshra Hussien, Specialist of Reproductive Health, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: boshahussien2021
Record Dates: First submitted 2023-10-15; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Complications of DMPA Injectable Contraceptives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women using DMPA after 6 weeks postpartum (Experimental)
  Interventions: Device: Depot-medroxy Progesterone Acetate Injectable Contraceptives
- Women using DMPA after 1 week postpartum (Experimental)
  Interventions: Device: Depot-medroxy Progesterone Acetate Injectable Contraceptives

INTERVENTIONS:
Device: Depot-medroxy Progesterone Acetate Injectable Contraceptives — Depot-medroxy progesterone acetate injectable contraceptives

SUMMARY:
This study aims to identify the effect of using Depot-medroxy progesterone acetate injectable contraceptives on lactating women mother and infant in 1st week versus 6th week postpartum initiation.

This study is open labeled -randomized clinical trial was used. It was conducted at woman's health hospital, Assuit University. This study applied on 120 lactating women, who divided into two equal group I (who used DMPA injectable in the 1st week postpartum) and group II (who used DMPA injectable in the 6th week postpartum). Each group included 60 lactating women). Follow up was carried out after 3 months from the first dose to determine the changes in the studied women's menstrual period, weight, breast feedings…etc.

ELIGIBILITY:
Inclusion Criteria:

Desire contraception for at least one year Apparently healthy participant Age 20- 40 years old Term delivery Birth weight >2.5 kg multipara Intend to breastfeed at time of hospital discharge Those delivered normally or by caesarean section Ready to follow and need immediate contraception

Exclusion Criteria:

Maternal health problems (DM, HTN, cardiac disease, anaemia, or any other obvious problem) Any maternal complications during labour Preterm delivery IUGR

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pattern of vaginal bleeding postpartum | 2021 to 2023
  Number of bleeding days- number of pads per day

SECONDARY OUTCOMES:
Duration and frequency of breast milk | 2021 to 2023
  score of frequency of breast feeding

CONTACTS AND LOCATIONS:
Locations (1):
- Boshra Hussien Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No